CLINICAL TRIAL: NCT01831505
Title: Feasibility of Assessing Lymphoma Response to Precise Local Injection of Candidate Chemotherapy Agents Using the CIVO(tm) Microdosing System
Brief Title: Feasibility of Assessing Lymphoma Response to Precise Local Injection of Candidate Chemotherapy Agents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Presage Biosciences (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRS-1; R42CA144104-02 (NIH)
Record Dates: First submitted 2013-04-08; First posted 2013-04-15 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Lymphoma
Keywords: personalized medicine; in vivo drug sensitivity; chemotherapy; lymphoma; microinjection
MeSH Terms: conditions — Lymphoma | interventions — Vincristine; Doxorubicin; Bendamustine Hydrochloride; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multiple drug microinjection (Experimental): Multiple drug microinjection with locally injected rituximab, vincristine, doxorubicin, bendamustine, prednisolone, or a combination of them
  Interventions: Drug: Multiple drug microinjection: rituximab, vincristine, doxorubicin, bendamustine, prednisolone or a combination of them

INTERVENTIONS:
Drug: Multiple drug microinjection: rituximab, vincristine, doxorubicin, bendamustine, prednisolone or a combination of them

SUMMARY:
Many cancer patients are prescribed drugs to which their cancer is already resistant - and thus suffer toxicity with no potential for benefit. Previous attempts to assess chemoresistance or sensitivity in vitro have failed. This is a feasibility study in human patients with newly diagnosed or recurrent lymphoma to determine how human cancerous lymph nodes in situ respond to standard of care therapeutics precisely microinjected with the CIVO(tm) microdosing system.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* Has enlarged lymph node(s) highly suspicious of lymphoma; or has been diagnosed with lymphoma but is untreated; or has persistent recurrent, or progressive lymphoma
* At least one enlarged lymph node that is considered accessible for percutaneous injection by the investigator and that is at least 2 cm in longest dimension.
* ECOG performance status of 0-2 (or a Karnofsky performance status of >50%).
* Labs required for enrollment: Absolute neutrophil count > 1000/mm3, platelet count > 50,000/mm3, hematocrit > 25%, creatinine <3.0 mg/dl, total bilirubin <4.0 mg/dl, SGOT and SGPT less than five times the institutional upper limits of normal.

Exclusion Criteria:

* Lymphoma patients in which the delay of surgery until the lymph node resection date or other factors associated with the study are not feasible.
* Patients with central nervous system disease.
* Any therapy that is potentially immunosuppressive or has anticancer activity in the 4 weeks prior to device microinjection.
* Patients with active fungal, viral, or bacterial infections
* Pregnant women.
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the response to locally injected drugs | 1-3 days post injection after injection

SECONDARY OUTCOMES:
Evaluate the safety profile of multiple simultaneous microinjections using custom syringe | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Oliver W Press, MD, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Seattle Cancer Care Alliance, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No